CLINICAL TRIAL: NCT03092206
Title: Changes in Insulin Sensitivity in Healthy Volunteers Taking Tenofovir Alafenamide (TAF)-Containing Antiretroviral Medication: The TAF-IR Study
Brief Title: Changes in Insulin Sensitivity in Healthy Volunteers Taking Tenofovir Alafenamide (TAF)-Containing Antiretroviral Medication
Acronym: TAF-IR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAF-1688-0030-I
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — emtricitabine tenofovir alafenamide; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Group 1: F/TAF ; oral; Dose: 25/200 mg; Frequency: QD Group 2: E/C/F/TAF; oral; Dose: 150/150/200/10 mg; Frequency: QD Group 3: R/F/TAF; oral; Dose: 25/200/25 mg; Frequency: QD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): F/TAF ; oral; Dose: 25/200 mg; Frequency: QD
  Interventions: Drug: F/TAF
- Group 2 (Experimental): Group 2: E/C/F/TAF; oral; Dose: 150/150/200/10 mg; Frequency: QD
  Interventions: Drug: E/C/F/TAF
- Group 3 (Experimental): Group 3: R/F/TAF; oral; Dose: 25/200/25 mg; Frequency: QD
  Interventions: Drug: R/F/TAF

INTERVENTIONS:
Drug: F/TAF — antiretroviral therapy
  Other Names: Descovy
  Arms: Group 1
Drug: E/C/F/TAF — antiretroviral therapy
  Other Names: Genvoya
  Arms: Group 2
Drug: R/F/TAF — antiretroviral therapy
  Other Names: Odefsey
  Arms: Group 3

SUMMARY:
Investigation of possible changes in insulin sensitivity in healthy volunteers taking the following HIV treatment combinations: F/TAF (group 1) as compared to E/C/F/TAF (group 2) as compared to R/F/TAF (group 3). The measurement of insulin sensitivity will be performed in 30 HIV-negative healthy non-obese (BMI 18-25) male volunteers before and after 14±2 days of treatment. The volunteers will be randomly assigned to one of the three groups. Changes in insulin sensitivity will be measured by golden standard hyperinsulinemic euglycemic clamp (HEGC) technique, using glucose and insulin infusion as diagnostic agents

DETAILED DESCRIPTION:
Nearly immediately following the characterization of HIV, the metabolic disturbances in HIV-positive patients, particularly changes in insulin sensitivity, were reported. The chronic inflammation due to metabolic changes caused by HIV-Infection on one hand and the antiretroviral therapy (ART) itself on the other hand were considered major contributors to pathological changes in insulin sensitivity in HIV-positive patients. There were two possible mechanisms discussed in the literature: Direct effects on insulin-associated cellular glucose uptake and indirect effects of changes in lipid metabolism, i.e. the lipotoxicity. Particularly, thymidine analogues, such as nucleoside reverse transcriptase inhibitors (NRTI) were strongly linked to lipotoxicity and depletion of mitochondric DNA, causing insulin resistance (IR) in HIV-positive patients and healthy volunteers, ultimately resulting in overt diabetes mellitus. Furthermore, protease inhibitors (PI) showed lipotoxicity, further increasing insulin resistance.

The incidence of insulin resistance and, ultimately, diabetes mellitus in patients receiving ART increases over time, significantly contributing to cardiovascular morbidity and mortality in HIV-positive patients. Due to significant increases both in life expectation and duration of ART in HIV-patients, the early recognition of unfavorable metabolic changes (i. e. insulin resistance) gains in importance. Particularly, the considerations of long-term toxicity and safety of ART are receiving more and more attention. Unfortunately, the appropriate strategies for screening, surveillance and therapeutic consequences are not well established in HIV-positive patients.

While the very well established HIV nucleoside reverse transcriptase inhibitor Tenofovir disaproxil fumarate (TDF) was associated with a favorable influence on lipids and with no known negative effects on insulin sensitivity, the new drug Tenofovir alafenamide (TAF) has not been analyzed in concern of changes in insulin sensitivity yet. As TAF has been recently submitted for approval by FDA and EMEA for treatment of HIV-positive patients, widespread use and potential replacement of TDF can be expected soon. Fixed dose combinations with Emtricitabine (F/TAF) or cobicistat-boosted elvitegravir (E/C/F/TAF) or rilpivirine (R/F/TAF) have been developed and will take part in ART settings. Unfortunately, only limited data exists on metabolic effects of TAF or TAF-containing fixed dose combination drugs, particularly concerning changes in lipid metabolism and insulin sensitivity in HIV-positive patients or healthy volunteers. For providing more safety data concerning changes in insulin sensitivity and associated effects on lipids more data should be provided.

We intend to investigate the possible changes in insulin sensitivity, measured as described below by "hyperinsulinemic eugylcemic clamp" in healthy volunteers taking TAF/FTC (group 1) as compared to E/C/F/TAF (group 2) as compared to R/F/TAF (group 3). To our best of knowledge, there are currently no data available investigating changes in insulin sensitivity of TAF-containing ART-regiments.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy volunteers, age range ≥18-40 years
* Written informed consent and willingness to attend study visits
* Willingness for taking study medication during study period
* Birth control during study period

Exclusion Criteria:

* Participation in other interventional clinical trials and/or participation in another clinical trial with medicinal products within the last 4 weeks
* Known allergies or contraindications against study medication
* Known metabolic dysfunction, e.g. Hypertriglyceridemia or Diabetes mellitus
* Smoking or alcohol abuse (> 15g/day alcohol consumption)
* Documented HIV-infection
* BMI <18 >25
* Recurrent medication or any antiretroviral medication within the last 30 days
* ALT, AST, Bilirubin, Creatinine, TSH, blood pressure, heart rate, QTc are out of normal range

  o Normal ranges for clinical chemistry are defined by local laboratory. For blood pressure normal range is defined as 100/60-140/90; for heart rate 60-100
* Known liver, kidney, heart, pulmonary, gastrointestinal, endocrinological, rheumathoid, neurological, psychiatric or metabolic diseases
* Any situation of which the sponsors sees relevant contraindication against study participation
* Imprisoned or situated people

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity | 14±2 days
  To assess changes in insulin sensitivity (mean glucose disposal rate normalized to body weight (MBW [mg glucose/min*kg]) in HIV-negative, healthy, non-obese (BMI 18-25) male volunteers following 14±2 days of treatment with group 1 or group 2 or group 3, as measured by HEGC.

SECONDARY OUTCOMES:
changes in insulin sensitivity | 14 +/-2 days
  To asses changes in insulin sensitivity as measured by mean glucose disposal rate normalized to body weight and steady-state insulin concentration (MBW/L [mg glucose/min kg UIU]) and normalized to body weight and steady-state glucose concentration (MCR [dL/min kg]), HOMA-IR, HOMA-, QUICKI and 1/QUICKI indices in HIV-negative, healthy, non-obese male volunteers following 14 +/-2 days of administration of IMP in group 1, 2 or 3.
lipid metabolism | 14±2 days
  Changes in lipid metabolism in HIV-negative, healthy, non-obese male volunteers following 14±2 days of administration of IMP in group 1, 2 or 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar (IZAR), Munich, Germany

IPD SHARING:
Plan to Share IPD: No